CLINICAL TRIAL: NCT04063150
Title: Immunogenicity of Intramuscular and Intradermal Inactivated Poliovirus Vaccine in Routine Immunization
Brief Title: Immunogenicity of Intramuscular and Intradermal IPV
Acronym: IM and ID IPV
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19058
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Poliomyelitis
Keywords: inactivated poliovirus vaccine; fractional inactivated poliovirus vaccine; intradermal; intramuscular
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- IPV at 14 weeks + 9 months (Active Comparator): Participants in this arm will receive full doses (0.5 mL) of IPV at 14 weeks and 9 months of age.
  Interventions: Biological: IPV
- IPV at 6 weeks + 9 months (Active Comparator): Participants in this arm will receive full doses (0.5 mL) of IPV at 6 weeks and 9 months of age.
  Interventions: Biological: IPV
- fIPV ID at 6 weeks + 14 weeks + 9 months (Active Comparator): Participants in this arm will receive intradermal fractional doses (0.1 mL) of IPV at 6 weeks, 14 weeks, and 9 months of age.
  Interventions: Biological: fIPV (0.1 mL) ID
- fIPV ID at 14 weeks + 9 months (Active Comparator): Participants in this arm will receive intradermal fractional doses (0.1 mL) of IPV at 14 weeks and 9 months of age.
  Interventions: Biological: fIPV (0.1 mL) ID
- fIPV IM at 6 weeks + 14 weeks + 9 months (Active Comparator): Participants in this arm will receive intramuscular fractional doses (0.1 mL) of IPV at 6 weeks, 14 weeks, and 9 months of age.
  Interventions: Biological: fIPV (0.1mL) IM
- fIPV 0.1mL IM at 14 weeks + 9 months (Active Comparator): Participants in this arm will receive intramuscular fractional doses (0.1 mL) of IPV at 14 weeks and 9 months of age.
  Interventions: Biological: fIPV (0.1mL) IM
- fIPV 0.2mL IM at 14 weeks + 9 months (Active Comparator): Participants in this arm will receive intramuscular fractional doses (0.2 mL) of IPV at 14 weeks and 9 months of age.
  Interventions: Biological: fIPV (0.2mL) IM

INTERVENTIONS:
Biological: fIPV (0.1 mL) ID — Fractional dose of inactivated poliovirus vaccine that protects against types 1, 2, and 3 (all polio serotypes). Given as a 0.1 milliliter (mL) dose (fractional) by intradermal (ID) injection in lieu of the full 0.5 mL dose.
  Arms: fIPV ID at 14 weeks + 9 months; fIPV ID at 6 weeks + 14 weeks + 9 months
Biological: fIPV (0.1mL) IM — Fractional dose of inactivated poliovirus vaccine that protects against types 1, 2, and 3 (all polio serotypes). Given as a 0.1 milliliter (mL) dose (fractional) by intramuscular (IM) injection in lieu of the full 0.5 mL dose.
  Arms: fIPV 0.1mL IM at 14 weeks + 9 months; fIPV IM at 6 weeks + 14 weeks + 9 months
Biological: fIPV (0.2mL) IM — Fractional dose of inactivated poliovirus vaccine that protects against types 1, 2, and 3 (all polio serotypes). Given as a 0.2 milliliter (mL) dose (fractional) by intramuscular (IM) injection in lieu of the full 0.5 mL dose.
  Arms: fIPV 0.2mL IM at 14 weeks + 9 months
Biological: IPV — Full dose of inactivated poliovirus vaccine that protects against types 1, 2, and 3 (all polio serotypes). Given as a 0.5 milliliter (mL) dose by intramuscular (IM) injection.
  Arms: IPV at 14 weeks + 9 months; IPV at 6 weeks + 9 months

SUMMARY:
This is an open-label phase IV randomized clinical trial that will compare immune responses among infants who receive different dose schedules of either fractional dose or full dose inactivated poliovirus vaccine (IPV), delivered either intramuscularly or intradermally.

Note: This study was terminated early due to the COVID-19 pandemic. Due to early study closure, the study objectives could not be evaluated as planned. Both of the primary objectives and several secondary objectives could not be evaluated because none of the study participants reached the corresponding endpoint. Due to limited sample size, the analysis approach for four secondary objectives was changed from a non-inferiority assessment to a comparison of proportions between groups.

DETAILED DESCRIPTION:
Oral poliovirus vaccine (OPV) cessation is essential to achieve eradication of polio as OPV contains live poliovirus, which can mutate and become neurovirulent. After OPV cessation, inactivated poliovirus vaccine (IPV) will be the only polio vaccine used for routine immunization. This clinical trial will provide poliovirus type-specific immunogenicity data on an IPV or fractional-dose IPV (fIPV)-only schedule for routine immunization, which will be important for post OPV cessation era. For fIPV, it will provide immunogenicity data on fIPV administered either intradermally (ID) or intramuscularly (IM) and allow a direct comparison of the two methods.

Healthy infants 6 weeks of age will be enrolled at two study clinics in Dhaka, Bangladesh, and randomized to one of seven study arms. Infants will be followed-up until 10 months of age through clinic visits. Blood specimens will be collected to test for immunological response.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants 6 weeks of age
* Parents that consent for participation in the full length of the study.
* Parents that are able to understand and comply with planned study procedures.

Exclusion Criteria:

* Parents and infants who are unable to participate in the full length of the study.
* A diagnosis or suspicion of immunodeficiency disorder either in the infant or in an immediate family member.
* A diagnosis or suspicion of bleeding disorder that would contraindicate parenteral administration of IPV or collection of blood by venipuncture.
* Acute diarrhoea, infection or illness at the time of enrolment (6 weeks of age) that would require infant's admission to a hospital.
* Acute vomiting and intolerance to liquids within 24 hours before the enrolment visit (6 weeks of age).
* Evidence of a chronic medical condition identified by a study medical officer during physical exam.
* Receipt of any polio vaccine (OPV or IPV) before enrolment based upon documentation or parental recall.
* Known allergy/sensitivity or reaction to polio vaccine, or its contents.
* Infants from multiple births. Infants from multiple births will be excluded because the infant(s) who is/are not enrolled would likely receive OPV through routine immunization and transmit vaccine poliovirus to the enrolled infant. Even if all births from a multiple birth could be enrolled in the study, we will exclude multiple births as discontinuation of one may lead to discontinuation of multiple participants.
* Infants from premature births (<37 weeks of gestation).

Ages: 42 Days to 48 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 958 (Actual)
Dates: Start 2019-10-06 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Vaccine response | Measured four weeks after administration of study vaccine(s).
  Dichotomous (yes/no) variable defined as participants who are either seronegative (<1:8 titers) at baseline who become seropositive (≥1:8) after vaccination (seroconversion) or participants who demonstrate a four-fold rise in titers after vaccination between two specimens, e.g. a change from 1:8 to 1:32, after adjusting for expected decay in maternal antibodies. Antibody titers at 6 weeks of age will be the starting point for the expected decline in maternal antibodies, assuming at half-life of 28 days.

SECONDARY OUTCOMES:
Reciprocal antibody titers | Measured four weeks after administration of study vaccine(s).
  Variable of the observed reciprocal antibody titer results.

CONTACTS AND LOCATIONS:
Locations (1):
- icddr,b study clinics (Mirpur and CTU Dhaka), Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No